CLINICAL TRIAL: NCT06332079
Title: Phase II Study Evaluating Holmium-166 TARE Followed by Maintenance Therapy in Liver Limited Unresectable Colorectal Cancer Patients After First-line Chemotherapy and Target Agents
Brief Title: Holmium-166 TARE in Liver Limited Unresectable Colorectal Cancer Patients
Acronym: HAITI
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Medical devices (QuiremScout/QuiremSpheres) no longer available due to discontinuation of production by the manufacturer
Sponsor: Gruppo Oncologico del Nord-Ovest (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HAITI 2023-505356-22-00
Record Dates: First submitted 2024-03-08; First posted 2024-03-27 (Actual); Last update posted 2026-01-05 (Actual); Status verified 2025-12

CONDITIONS: Colorectal Cancer Metastatic
Keywords: HOLMIUM; TARE; Maintenance therapy; Liver-limited colorectal cancer; Unresectable colorectal cancer
MeSH Terms: interventions — Cetuximab; Panitumumab; Fluorouracil; Bevacizumab; Capecitabine

STUDY DESIGN:
Intervention Model Description: Two cohorts of patients will be included according to the two main prognostic populations in mCRC (left sided, RAS/BRAF wild-type and, right-sided and/or RAS mutated tumors) treated with different maintenance therapy (fluoropyrimidine plus anti-EGFR or bevacizumab).
  A total of 23 patients will be enrolled in each cohort.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- COHORT A/B (Experimental): Eligible patients will receive Scout dose procedure. After 1-2 weeks, patients eligible for radioembolization will receive 166Ho-TARE and at least after 3 weeks, maintenance treatment with fluoropyrimidine plus target agents (anti-EGFR or bevacizumab) according to the respective study cohort.
  Maintenance treatment:
  Cohort A:
  * CETUXIMAB iv day1, over 1 hours, 500 mg/sqm or PANITUMUMAB iv over 1 hours, 6 mg/kg, every 14 days
  * LED 200 mg/sqm iv over 1 hour, day 1
  * 5-FLUOROURACIL ic 48 h, starting on day 1 every 14 days; 2400 mg/sqm and 400 mg/sqm bolus if FOLFOX/FOLFIRI in the induction treatment
  Cohort B:
  * BEVACIZUMAB 5 mg/kg iv biweekly day1, over 30 minutes
  * LED 200 mg/sqm iv over 1 hour, day 1
  * 5-FLUOROURACIL ic 48 h, starting on day 1 every 14 days; 2400 mg/sqm and 400 mg/sqm bolus if FOLFOX/FOLFIRI in the induction treatment
  CAPECITABINE, 1000 mg/sqm orally twice daily, day 1-14, plus bevacizumab 7,5 mg/kg iv every 21 days is allowed.
  Interventions: Procedure: 166Holmium TARE; Drug: Cetuximab; Drug: Panitumumab; Drug: 5-Fluorouracil; Drug: Bevacizumab; Drug: Capecitabine

INTERVENTIONS:
Procedure: 166Holmium TARE — 166Ho-TARE treatment comprises of two hospital visits: one for a work-up procedure and another for the therapy procedure, with usually a 1-2 weeks interval.
Drug: Cetuximab — Target agent
Drug: Panitumumab — Target agent
Drug: 5-Fluorouracil — Chemotherapy
Drug: Bevacizumab — Target agent
Drug: Capecitabine — Chemotherapy

SUMMARY:
The aim of this study is to assess the efficacy of 166Ho-TARE followed by maintenance therapy with fluoropyrimidine and anti-EGFR or bevacizumab in liver-limited unresectable colorectal cancer patients, in terms of progression free rate 9- and 8-months for cohort A and B, respectively.

DETAILED DESCRIPTION:
HAITI is a phase II, single-arm trial of 166Ho-TARE followed by maintenance therapy in liver-limited unresectable colorectal cancer patients, achieving partial response or stable disease according to RECIST 1.1 criteria after 6-12 cycles of induction first-line chemotherapy.

Two cohorts of patients are included:

* left sided RAS/BRAF wild-type (cohort A)
* right-sided and/or RAS mutated (cohort B)

Enrolled patients will be treated with different maintenance therapy according to study cohort (fluoropyrimidine + anti-EGFR or bevacizumab).

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent to study procedures;
* Age ≥18 years;
* Histologically proven diagnosis of colorectal adenocarcinoma, with or without primary tumour in situ;
* Liver-only disease at radiological exams involving less than 50% of liver volume;
* Eastern Cooperative Oncology Group Performance Status (ECOG PS) ≤2;
* Patients with partial response or stable disease according to RECIST 1.1 criteria deemed unresectable after 6-12 cycles of induction first-line chemotherapy;
* Life expectancy of at least 12 weeks;
* Hematopoietic function: absolute neutrophil count ≥ 1,500/mm3; platelet count

  ≥100,000/mm3; haemoglobin level ≥ 9 g/dL;
* Liver function: total bilirubin ≤ 1.5 times upper limit of normal (ULN); alkaline phosphatase

  ≤ 5 times ULN; AST ≤ 5 times ULN;
* Renal function: creatinine clearance > 50 mL/min or serum creatinine 1.5 x UNL; no renal disease that would preclude study treatment or follow-up;
* Women of childbearing potential must have a negative blood pregnancy test at the screening visit. For this trial, women of childbearing potential are defined as all women after puberty, unless they are postmenopausal for at least 12 months, are surgically sterile, or are sexually inactive. A postmenopausal state is defined as no menses for 12 months without an alternative medical cause. A high follicle stimulating hormone (FSH) level in the postmenopausal range may be used to confirm a post-menopausal state in women not using hormonal contraception or hormonal replacement therapy. However, in the absence of 12 months of amenorrhea, a single FSH measurement is insufficient;
* Subjects and their partners must be willing to avoid pregnancy during the trial. Male subjects with female partners of childbearing potential and female subjects of childbearing potential must, therefore, be willing to use adequate contraception as outlined in Section 7.5 - Contraception, starting during study screening visit throughout the study period up to 180 days after the last dose of chemotherapy Note: Abstinence is acceptable if this is the usual lifestyle and preferred contraception for the subject;
* Will and ability to comply with the protocol

Inclusion criteria for Cohort A:

* RAS/BRAF wild-type and left sided primary tumor
* First-line induction chemotherapy regimen permitted up to 6-12 cycles with:

FOLFOX or FOLFIRI + anti-EGFR (cetuximab or panitumumab). Patients who interrupted anti-EGFR target therapy during induction phase due to toxicity or other reasons, candidate to maintenance with fluoropyridine alone therapy can be enrolled.

Inclusion criteria for Cohort B:

* RAS mutated and/or right-sided primary tumor
* First-line induction chemotherapy regimen admitted up to 6-12 cycles with:

FOLFOX/FOLFIRI/XELOX + bevacizumab or FOLFOXIRI + bevacizumab. Patients who interrupted bevacizumab during induction phase due to toxicity or other reasons, candidate to maintenance with fluoropyridine alone therapy can be enrolled.

Exclusion Criteria:

* Patients with radiological evidence of extra liver distant metastases.
* Evidence of ascites, cirrhosis, portal hypertension, main portal venous tumour involvement or thrombosis, or any other contraindications to radioembolization treatment;
* Previous radiotherapy delivered to the liver;
* Patients with BRAF mutated and/or MSI-high tumours;
* Previous history of malignancy within the last 5 years will be excluded with the exception of localized basal and squamous cell carcinoma or cervical cancer in situ;
* Treatment with any investigational drug within 30 days prior to enrolment or 2 investigational agent half-lives (whichever is longer);
* Active uncontrolled infections or other clinically relevant concomitant illness contraindicating study procedures and treatment administration Clinically significant (e.g. active) cardiovascular disease for example cerebrovascular accidents (≤6 months), myocardial infarction (≤6 months), unstable angina, New York Heart Association (NYHA) grade II or greater congestive heart failure (CHF), serious cardiac arrhythmia requiring medication
* Pregnant or lactating women. Women of childbearing potential with either a positive or no pregnancy test at baseline. Sexually active males and females (of childbearing potential) unwilling to practice contraception during the study and until 180 days after the last trial treatment;
* History of a previous allergic reaction to contrast media that would preclude safe angiography of the hepatic arteries, in the opinion of the treating Interventional Radiologist;
* Known hypersensitivity to fluoropyrimidine, anti-VEGF or anti-EGFR MoAb.
* Psychiatric or addictive disorders, or other conditions that, in the opinion of the investigator, would preclude study participation;
* Withdrawal of the consent to take part to the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2024-03-13 (Actual); Primary Completion 2025-12-16 (Actual); Study Completion 2025-12-16 (Actual)

PRIMARY OUTCOMES:
Progression-free survival (PFS) Rate | 36 months
  PFS is defined as the time from study enrolment to the first documentation of objective disease progression or death due to any cause, whichever occurs first. PFS will be censored on the date of the last evaluable on study tumor assessment documenting absence of progressive disease for patients who are alive, on study and progression free at the time of the analysis.

SECONDARY OUTCOMES:
Overall Toxicity rate | 36 months
  Overall Toxicity rate is defined as the percentage of patients, relative to the total of enrolled subjects, who receive 166Ho-TARE and at least one cycle of chemotherapy, experiencing any adverse event, according to National Cancer Institute Common Toxicity Criteria (version 5.0) during the study treatment.
Grade 3/ Grade 4 Toxicity rate | 36 months
  Grade 3/ Grade 4 Toxicity rate is defined as the percentage of patients, relative to the total of enrolled subjects, who receive 166Ho-TARE and at least one cycle of chemotherapy, experiencing a specific adverse event of severity grade 3/ grade 4, according to National Cancer Institute Common Toxicity Criteria (version 5.0) during the study treatment.
Post-treatment Disease Control Rate (DCR) | 36 months
  Post-treatment DCR, is defined as the percentage of patients, relative to the total of enrolled subjects, achieving a complete (CR), partial (PR) response or stable disease (SD), according to RECIST 1.1 criteria, during the study treatment. The determination of clinical response will be based on investigator reported measurements. Tumor re-assessment with CT scan will be repeated every 8- weeks.
Progression free survival | 36 months
  Progression free survival (PFS), is defined as the time from study enrolment to the first documentation of objective disease progression or death due to any cause, whichever occurs first. PFS will be censored on the date of the last evaluable on study tumor assessment documenting absence of progressive disease for patients who are alive, on study and progression free at the time of the analysis.
Overall Survival | 36 months
  Overall Survival (OS), is defined as the time from enrolment to death from any cause. For patients still alive at the time of analysis, the OS time will be censored on the last date the patients were known to be alive.
Dose-response relationships | 36 months
  Dose-response relationships are defined as the relationships between the tumor-absorbed doses calculated on post-treatment SPECT-CT (dependent variables) and the following independent variables: tumor response (SD, PR, CR according to RECIST CRITERIA v 1.1), progression free survival rate, and Overall Survival.
Quality of Life (QoL) assessed using the EORTC QLQ-CR29 questionnaire | 36 months
  The EORTC QLQ-CR29 is a patient-reported outcome measure to evaluate health-related quality of life among colorectal cancer patients in research and clinical practice.
  QoL assessed using the EORTC QLQ-CR29 questionnaire will be evaluate at specific time-points (baseline, tumor reassessment and disease progression) and will be assessed through descriptive summary statistics.
Quality of Life (QoL) assessed using the EORTC QLQ-CR30 questionnaire | 36 months
  The EORTC QLQ-CR30 is 30-item instrument designed to measure quality of life in all cancer patients.
  QoL assessed using the EORTC QLQ-CR30 questionnaire will be evaluate at specific time-points (baseline, tumor reassessment and disease progression) and will be assessed through descriptive summary statistics.
Quality of Life (QoL) assessed using the EuroQol EQ-5D questionnaire | 36 months
  The EuroQol EQ-5D comprises five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems and extreme problems.
  QoL assessed using the EuroQol EQ-5D questionnaire will be evaluate at specific time-points (baseline, tumor reassessment and disease progression) and will be assessed through descriptive summary statistics.

CONTACTS AND LOCATIONS:
Overall Officials: Gianluca Masi, MD, Principal Investigator — Azienda Ospedaliero, Universitaria Pisana
Locations (1):
- Azienda Ospedaliero Universitaria Pisana, Pisa, Italy

IPD SHARING:
Plan to Share IPD: No